CLINICAL TRIAL: NCT01649661
Title: Epidemiology of MRI Parenchymal Enhancement: A New Marker of Breast Cancer Risk
Brief Title: MRI Parenchymal Enhancement: A New Marker of Breast Cancer Risk
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); University of Southern California (Other); University of Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 12-125
Record Dates: First submitted 2012-07-19; First posted 2012-07-25 (Estimated); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Cancer Free Women
Keywords: MRI; 12-125; premenopausal women; postmenopausal women; questionnaire
MeSH Terms: interventions — Surveys and Questionnaires; Health Records, Personal; Reproductive History; Ethanol; Smoking Devices

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sample collected at time of MRI for serum hormone analysis Postmenopausal women only

GROUPS / COHORTS (2):
- premenopausal women: Only women already scheduled for a breast MRI will be included in the study, no additional MRIs will be scheduled for study purposes.
  Interventions: Behavioral: questionnaire
- postmenopausal women: Only women already scheduled for a breast MRI will be included in the study, no additional MRIs will be scheduled for study purposes.
  Interventions: Behavioral: questionnaire

INTERVENTIONS:
Behavioral: questionnaire
  Other Names: The study questionnaire is a 15-20 minute survey at or shortly after the time of MRI consisting of 27; questions in 7 domains:background information (e.g., date of birth, country of birth, race/ethnicity), medical; history, family history of cancer, reproductive history, use of hormonal medications, alcohol and; smoking, contact information/comments.

SUMMARY:
The purpose of this study is to learn about how a woman's health history influences what a normal breast looks like on an MRI. The investigators also want to learn about how the amount of different natural hormones a woman has affects how the breast looks on an MRI. The investigator's hope is that this will help to find women at a high-risk of breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* age 21 years or older
* be a cancer-free pre- or postmenopausal woman
* have no prior personal history of any cancer (including DCIS, excluding nonmelanoma skin-cancer)
* able to speak and read English because the questionnaire is only available in English
* able to provide informed consent

Exclusion Criteria:

* are pregnant at the time of MRI
* have a prior personal history of any cancer (including DCIS, excluding nonmelanoma skin cancer)

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The proposed study will involve cancer-free women who are undergoing breast MRI screening at MSKCC.
Sampling Method: Non-Probability Sample
Enrollment: 437 (Actual)
Dates: Start 2012-07; Primary Completion 2023-01-25 (Actual); Study Completion 2023-01-25 (Actual)

PRIMARY OUTCOMES:
breast cancer risk factors and background parenchymal enhancement (BPE). | 1 year
  A comparison of the distribution of breast cancer risk factors in women with low and high levels of BPE. The relationship between risk factors and categories of BPE (minimal/mild/moderate/marked) will be determined using ordinal logistic regression.

SECONDARY OUTCOMES:
relationship between BPE and serum hormone levels at the time of MRI | 1 year
  Determine the relationship between serum hormone levels (testosterone, estradiol (E2), estrone (E1), androstenedione (A4) and sex hormone binding globulin (SHBG)) at the time of MRI and degree of BPE in healthy high-risk postmenopausal women. The association between circulating serum hormone levels and BPE will be determined using linear regression.

CONTACTS AND LOCATIONS:
Overall Officials: Janice Sung, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/